CLINICAL TRIAL: NCT06997666
Title: The Effect of Prone Position on Oxygen Saturation, Blood Gas Parameters, and Respiratory Rate in Intensive Care Patients With COVID-19-induced ARDS
Brief Title: Effect of Prone Position on Oxygen, Blood Gas, and Respiratory Parameters in Intensive Care Patients With COVID-19-induced ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medet Korkmaz (Other)
Responsible Party: Sponsor-Investigator, Medet Korkmaz, professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 626
Record Dates: First submitted 2025-05-26; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: COVID - 19; ARDS (Acute Respiratory Distress Syndrome)
Keywords: ARDS; COVID-19; Nursing; Blood gas values; Prone position
MeSH Terms: conditions — COVID-19; Acute Lung Injury | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Position Group (Experimental): Patients in this group were placed in the prone position for 30 minutes once daily on two consecutive days. Oxygen saturation (SpO₂), blood gas parameters (SaO₂, PO₂, PCO₂, pH, lactate, sodium), and respiratory rate were measured before and after the intervention. No other treatment was altered.
  Interventions: Procedure: Prone Position
- Supine Standard Care Group (No Intervention): Patients in this group received standard intensive care in the supine position. No additional interventions were applied. Oxygen saturation (SpO₂), blood gas parameters (SaO₂, PO₂, PCO₂, pH, lactate, sodium), and respiratory rate were measured at the same intervals as the intervention group.

INTERVENTIONS:
Procedure: Prone Position — Patients assigned to the Prone Position Group were placed in the prone position (lying face down) for 30 minutes once daily over two consecutive days while hospitalized in the ICU for COVID-19-induced ARDS. The intervention was performed between 12:30 and 13:00 under nurse supervision. Oxygen saturation, blood gas parameters (SaO₂, PO₂, PCO₂, pH, lactate, sodium), and respiratory rate were measured before and after each prone positioning session. The procedure was standardized across patients and no additional treatments were introduced during the intervention period.
  Arms: Prone Position Group

SUMMARY:
This randomized controlled trial aimed to investigate the effect of the prone position on oxygen saturation, arterial blood gas parameters, and respiratory rate in intensive care patients diagnosed with COVID-19-induced Acute Respiratory Distress Syndrome (ARDS). A total of 90 patients (45 in the prone positioning group and 45 in the control group) were included. The intervention group received a 30-minute prone positioning procedure, while the control group received standard ICU care. Data were collected using a Demographic Information Form and clinical monitoring of respiratory and blood gas parameters across six time points over two days.

DETAILED DESCRIPTION:
This randomized controlled trial investigated the short-term physiological effects of prone positioning in intubated intensive care patients diagnosed with COVID-19-induced Acute Respiratory Distress Syndrome (ARDS). A total of 90 patients were included, with 45 in the experimental group and 45 in the control group. Patients in the experimental group were placed in the prone position for 30 minutes on two consecutive days, while the control group received standard ICU care without prone positioning.

Oxygen saturation (SpO₂, SaO₂), arterial blood gas parameters (PO₂, PCO₂, pH, lactate, sodium), and respiratory rate were measured at six time points to evaluate the effectiveness of the intervention. The study was conducted in the general and intermediate intensive care units of a public hospital in eastern Turkey, which was designated as a COVID-19 treatment center during the pandemic.

The study's primary objective was to determine whether prone positioning could improve oxygenation and respiratory efficiency in critically ill patients with COVID-19-related ARDS. Secondary outcomes included changes in blood gas and metabolic parameters. The results suggested that prone positioning had a beneficial impact on oxygen saturation and respiratory rate without causing adverse changes in blood gas chemistry. The study was ethically approved and conducted in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Admission to an intensive care unit (ICU)
* Confirmed diagnosis of COVID-19
* Developed Acute Respiratory Distress Syndrome (ARDS) due to COVID-19
* Intubated at the time of enrollment
* Provided informed verbal and written consent (or consent provided by legal representative)

Exclusion Criteria:

* Significant hearing or vision impairments affecting communication
* Cognitive impairment or inability to understand instructions
* Patient died during the course of the study
* Early discharge from intensive care before completion of all measurements
* Non-intubated patients whose level of consciousness could not be monitored

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen Saturation (SpO₂) | Baseline and six repeated measurements over two consecutive days
  Measurement of arterial oxygen saturation (SaO₂), partial pressure of oxygen (PO₂), partial pressure of carbon dioxide (PCO₂), and pH from blood gas analysis to assess respiratory and metabolic effects of prone positioning.

SECONDARY OUTCOMES:
Change in Arterial Blood Gas Parameters (SaO₂, PO₂, PCO₂, pH) | Baseline and six repeated measurements over two consecutive days
  Measurement of arterial oxygen saturation (SaO₂), partial pressure of oxygen (PO₂), partial pressure of carbon dioxide (PCO₂), and pH from blood gas analysis to assess respiratory and metabolic effects of prone positioning.

OTHER OUTCOMES:
Change in Respiratory Rate | Baseline and six repeated measurements over two consecutive days
  Monitoring of respiratory rate (breaths per minute) before and after prone positioning to assess its impact on breathing efficiency.
Change in Serum Lactate and Sodium Levels | Baseline and six repeated measurements over two consecutive days
  Assessment of serum lactate and sodium concentrations to identify any metabolic changes associated with prone positioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Diyarbakır Provincial Health Directorate, 21000, Diyarbakır, Turkey, Diyarbakır, Turkey (Türkiye)

REFERENCES:
- [Derived] Tekin V, Korkmaz M. The effect of prone position on oxygen saturation, blood gas parameters, and respiratory rate in intensive care patients with COVID-19-induced ARDS. Sci Rep. 2025 Nov 29;16(1):108. doi: 10.1038/s41598-025-28844-3. PMID 41318642

DOCUMENTS (3):
  • Study Protocol (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT06997666/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT06997666/SAP_001.pdf
  • Informed Consent Form (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT06997666/ICF_002.pdf